CLINICAL TRIAL: NCT05255536
Title: The Effect of Different Local Anesthetic Volumes of Serratus Anterior Plan Block Performed With Ultrasound on Acute Pain After Video-Assisted Thoracoscopic Surgery
Brief Title: Effect of Different Local Anesthetic Volumes of Serratus Anterior Plan Block After Video-Assisted Thoracoscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.Kurul-E1-22-2371
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Serratus Anterior Plane Block; Pain, Postoperative; Thoracic Surgery, Video-Assisted; Local Anesthetic
MeSH Terms: conditions — Pain, Postoperative | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Anterior Plan Block with 20 ml %0.25 Bupivacaine (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle will be advanced via the in-plane technique above the serratus anterior muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 20 ml 0.25% bupivacaine will be injected into the area.
  Interventions: Procedure: Serratus Anterior Plan Block with 20 ml
- Serratus Anterior Plan Block with 30 ml %0.25 Bupivacaine (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle will be advanced via the in-plane technique above the serratus anterior muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 30 ml 0.25% bupivacaine will be injected into the area.
  Interventions: Procedure: Serratus Anterior Plan Block with 30 ml

INTERVENTIONS:
Procedure: Serratus Anterior Plan Block with 20 ml — Superficial serratus anterior plane block with 20 ml will be applied to the patients under real-time ultrasound guidance.
  Other Names: Drug
  Arms: Serratus Anterior Plan Block with 20 ml %0.25 Bupivacaine
Procedure: Serratus Anterior Plan Block with 30 ml — Superficial serratus anterior plane block with 30 ml will be applied to the patients under real-time ultrasound guidance.
  Other Names: Drug
  Arms: Serratus Anterior Plan Block with 30 ml %0.25 Bupivacaine

SUMMARY:
Video-assisted thoracic surgery (VATS) has become a common procedure in thoracic surgery. Severe postoperative pain may be encountered in patients undergoing VATS. Analgesic methods such as thoracic paravertebral block (TPVB), intercostal block, serratus anterior plane block (SAPB), and erector spinae plane block (ESPB) are widely used for VATS. Among these methods, ultrasound (US) guided TPVB is the most preferred method. In recent years, the frequency of application of plane blocks as a component of multimodal analgesia has been increased. ESPB and SAPB are some of them. In addition, SAPB application is increasing in patients who underwent thoracotomy and VATS. There is no consensus on the dose of analgesia in these studies. There are studies on volumes between 10 ml and 40 ml in the literature. In this study, it was aimed to compare the volumes of 20 ml and 30 ml containing local anesthetic at the same concentration (0.25% bupivacaine) of SAPB block to be performed with USG in patients who underwent VATS.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* ASA physical status I-II-III
* BMI 18 to 30 kg/m2
* Elective video assisted thoracoscopic surgery

Exclusion Criteria:

* Patient refusing the procedure
* Emergency surgery
* Chronic opioid or analgesic use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | 48 hours after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 1st, 2nd, 4th, 8th, 16th, 24th and 48th hours after surgery.

SECONDARY OUTCOMES:
Morphine Consumption | 24 hours after surgery
  Morphine consumption for 24 hours will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Musa Zengin, MD, Principal Investigator — Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)